CLINICAL TRIAL: NCT01621542
Title: Initial Phase 1 Study of WT2725 in Patients With Advanced Malignancies
Brief Title: Clinical Study of WT2725 in Patients With Advanced Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Collaborators: Sumitomo Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D8350004
Record Dates: First submitted 2012-06-06; First posted 2012-06-18 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2019-07-17 (Actual); Status verified 2019-05

CONDITIONS: Cancer
Keywords: Cancer; Vaccine; Oncology; Malignancies; Wilms' Tumor; WT1; Ovarian; Glioblastoma [GBM]; Acute myeloid leukemia [AML]
MeSH Terms: conditions — Neoplasms; Wilms Tumor; Leukemia, Myeloid, Acute

STUDY DESIGN:
Masking Description: Open label
Oversight: Data Monitoring Committee: No

ARMS (1):
- WT2725 (Experimental): WT2725; injection
  Interventions: Biological: WT2725

INTERVENTIONS:
Biological: WT2725 — WT2725 injection Study drug will be administered every 1-4 weeks

SUMMARY:
This clinical study is designed to evaluate the safety, immunogenicity and antitumor activity of WT2725. WT2725 will be administered to patients with advanced malignancies known to overexpress WT1

DETAILED DESCRIPTION:
Treatment with other WT1 vaccines in clinical trials has shown evidence of immunogenicity and clinical response in various malignancies.

This study will assist with determining which dose level(s) to use in future clinical studies and will evaluate both clinical and immunological response.

ELIGIBILITY:
Part 1 Inclusion Criteria:

* Patient must have an Eastern Cooperative Oncology Group (ECOG) Performance Score of 0, 1, or 2
* Patient must have one of the following histologically or cytologically documented measurable (may be measureable by tumor markers only, such as quantitative RT-PCR for WT1 transcript for AML, or CA-125 for ovarian carcinoma) advanced stage malignancies: non-small cell lung, ovarian, glioblastoma, and AML (not including acute promyelocytic leukemia), known to overexpress the WT1 protein.
* Patient must qualify with a study specific HLA typing assay.
* Haematological parameters:

  * Absolute neutrophil count (ANC) ≥ 1,000/μl
  * Platelet count ≥ 10.0x10(to the 4th power)/μl (≥ 5.0 x 10(to 4th power)/μl after stem cell transplant)
  * Hemoglobin ≥ 9.0 g/dL
  * Absolute lymphocyte count (ALC) ≥ 1,000/μl (≥ 500/μl after stem cell transplant) Note: After completion of dose escalation, patients with AML are not required to meet these hematologic criteria.
* Biochemical Parameters:

  * serum creatinine of ≤ 1.5x upper limit of normal (ULN) for the reference lab.
  * total bilirubin of ≤ 2.0 mg/dl (≤ 3.0 mg/dl for patients with known Gilbert's syndrome)
  * alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 3 times the ULN for the reference lab
* Patient must have access to archival tumor tissue sample or agree to undergo biopsy after study eligibility has been confirmed to obtain fresh sample for evaluation of WT1 expression. In place of archival tumor tissue samples, subjects with AML should have available a bone marrow aspirate and/or, bone marrow biopsy, with PCR for WT1 transcript performed before the first dose of study drug.

Note: The archived tumor tissue sample does not need to be delivered to the clinical site prior to enrollment of the patient, however its availability should be confirmed through provision of the accession number or other identification number.

Patient Inclusion Criteria - Part 2:

* Patient or his or her legal representatives must give written informed consent and privacy authorization prior to participation in the study.
* Patient must be willing and able to comply with the study procedures and visit schedules and must be able to follow verbal and written instructions.
* Patient must be ≥ 18 years of age.
* Women of childbearing potential and men with female sexual partners of childbearing potential must agree to abstain from sexual intercourse or use a double barrier method to determine if a woman is of childbearing potential (http://www.nccn.org/professionals/physician_gls/f_guidelines.asp).
* Patient must have an ECOG Performance Score of 0, 1, or 2 (refer to Appendix II).
* Patient has a life expectancy of at least 4 months.
* Patient must have histologically or cytologically documented measurable (may be measurable by tumor markers only, such as quantitative RT-PCR for WT1 transcript for AML) advanced stage glioblastoma or AML (not including acute promyelocytic leukemia), known to overexpress the WT1 protein. Note: Determination of WT1 expression will not be assessed prior to patient enrollment.
* Patient must have an advanced stage malignancy defined as meeting at least one of the following criteria:
* progressed or recurred despite standard therapy
* no standard therapy exists
* patient is intolerant of standard therapy
* patient is not a candidate for standard therapy
* Patient must be HLA-A*0201+ and/or HLA-A*0206+
* Patient with glioblastoma must have adequate bone marrow and immune reserve, as documented by:
* ANC ≥ 1000/μl (≥ 500/μl after stem cell transplant)
* Platelet count ≥ 10.0 x 1(to the 4th power)/μl (≥ 5.0 x 10(to the 4th power)/μl after stem cell transplant)
* Hemoglobin ≥ 9.0 g/dL
* ALC ≥ 900/μl (Note: Patients with AML are not required to meet these hematologic criteria).
* Patient must have adequate renal function documented by a serum creatinine of ≤ 1.5 times the ULN for the reference lab.
* Patient must have adequate hepatic function documented by a total bilirubin of ≤ 2.0 mg/dl (≤ 3.0 mg/dl for patients with known Gilbert's syndrome) and ALT and AST ≤ 3 times the ULN for the reference lab.
* Patient must have access to archival tumor tissue sample or agree to undergo biopsy after study eligibility has been confirmed to obtain fresh sample for evaluation of WT1 expression. In place of archival tumor tissue samples, patients with AML should have available a bone marrow aspirate and/or bone marrow biopsy with PCR for WT1 transcript performed before the first dose of study drug.

Note: The archived tumor tissue sample does not need to be delivered to the clinical site prior to enrollment of the patient, however its availability should be confirmed through provision of the accession number or other identification number.

• Patients with AML must be willing to undergo bone marrow aspiration/biopsy during treatment if there are no other indicators of measureable disease.

Part 1 Exclusion Criteria:

* Patient with an extensively disseminated primary glioblastoma.
* Patient with symptomatic brain metastases, ie, not neurologically stable or requiring treatment with corticosteroids, or central nervous system (CNS) leukemia.
* Patient with an infection requiring treatment with systemic antibiotics or antiviral medication or has completed treatment for such an infection within 4 days prior to planned initial dose of WT2725.
* Patient requiring systemic, pharmacologic doses of corticosteroids (equivalent to > 60 mg hydrocortisone/day or 2 mg dexamethasone/day). Replacement doses (equivalent to ≤ 5 mg prednisone/day), and topical, ophthalmic, and inhalation steroids are permitted as needed.
* Patient has a positive test for Hepatitis B surface antigen, Hepatitis C antibody, human immunodeficiency virus (HIV)-1, or HIV-2 antibody, or has a history of a positive result.
* Patient has received any of the following treatments within the specified timeframe prior to dosing:

  * endocrine therapy, immunotherapy, transfusion, hematopoietic factors within 14 days prior to planned first dose of study drug (Note: After completion of dose escalation, patients with AML are not required to meet these hematologic criteria, eg. transfusions and hematopoietic growth factors.)
  * chemotherapy including molecular-targeting therapy within 21 days (for molecular-targeted agents that are not associated with myelosuppression or immunosuppression, the minimum interval is 5 half-lives if that is less than 21 days)
  * surgery, radiation, or immunosuppressants within 28 days
  * investigational drug within 28 days
  * mitomycin-C or nitrosoureas within 42 days
* Patient with an unresolved ≥ Grade 2 AE from a previous antineoplastic treatment, excluding alopecia.
* Pregnant or lactating women
* Patient with an autoimmune condition
* Patients with serious unstable medical illness
* Patient with pleural effusion, ascites, or pericardial fluid requiring drainage.
* Patient is a staff member of the sponsor or clinical site and is involved in the conduct of the study or the relative of such a staff member.

Patient Exclusion Criteria - Part 2:

* Patient has an extensively disseminated primary glioblastoma.
* Patient has symptomatic brain metastases, ie, presence of neurological symptoms or requiring treatment with corticosteroids, or CNS leukemia.
* Patient has an infection and has had a body temperature of > 38.3˚C within 48 hours prior to planned first dose of study drug.
* Patient requires systemic, pharmacologic doses of corticosteroids (equivalent to > 60 mg hydrocortisone/day or 2 mg dexamethasone/day). Replacement doses (equivalent to ≤ 5 mg prednisone/day), and topical, ophthalmic, and inhalation steroids are permitted as needed.
* Patient has a positive test for Hepatitis B surface antigen, Hepatitis C antibody, HIV-1, or HIV-2 antibody, or has a history of a positive result.
* Patient has received any of the following treatments within the specified timeframe:

  * endocrine therapy, immunotherapy, transfusion, or hematopoietic factors within 14 days prior to planned first dose of study drug (Note: Patients with AML are not required to meet these hematologic criteria, eg, transfusions and hematopoietic growth factors.),
  * chemotherapy including molecular-targeting therapy within 21 days prior to planned first dose of study drug (for molecular-targeted agents that are notis 5 half-lives if that is less than 21 days),
  * surgery, radiation, or immunosuppressants within 28 days prior to planned first dose of study drug,
  * investigational drug within the 28 days prior to planned first dose of study drug, or
  * mitomycin-C or nitrosoureas within 42 days prior to planned first dose of study drug.

Note: Patients receiving LHRH agonists or antagonists or antiestrogens or aromatase inhibitors started and at a stable dose for at least 90 days prior to planned first dose of study drug are eligible. Patients are permitted one 28 day cycle of concurrent treatment with hydroxyurea during the study.

* Patient has an unresolved ≥ Grade 2 AE from a previous antineoplastic treatment, excluding alopecia.
* Woman who is pregnant or lactating or has a positive pregnancy test at screening. If a woman has a positive pregnancy test, further evaluation may be conducted to rule out ongoing pregnancy to allow the patient to be eligible.
* Patient has an autoimmune condition, including, but not limited to, multiple sclerosis, Grave's disease, vasculitis, systemic lupus erythematosus, rheumatoid arthritis, systemic sclerosis, myasthenia gravis, ankylosing spondylitis, Wegener's granulomatosis, ulcerative colitis, Crohn's disease, psoriasis requiring systemic therapy, pemphigus, temporal arteritis, dermatomyositis, Sjögren's syndrome, Goodpasture's syndrome, interstitial pneumonitis, interstitial nephritis, or Henoch-Schönlein purpura.
* Patient has in the opinion of the investigator any intercurrent conditions that could preclude their participation in the study, pose an undue medical hazard, or that could interfere with the interpretation of the study results, including, but not limited to, patients with congestive heart failure (NYHA Class III or IV; refer to Appendix III), unstable angina, cardiac arrhythmia requiring treatment, recent (within the prior 6 months) myocardial infarction, acute coronary syndrome or stroke, severe obstructive pulmonary disease, hypertension requiring more than2 medications for adequate control, or diabetes mellitus with more than 2 episodes of ketoacidosis in the prior 12 months.
* Patient has pleural effusion, ascites, or pericardial fluid requiring drainage. Note: Patient who had drain removal ≥ 14 days prior to planned first dose of study drug and has no sign of worsening is eligible.
* Patient has any other medical, psychiatric, or social condition, including substance abuse that in the opinion of the investigator would preclude participation in the study.
* Patient has had previous treatment with the study drug or other WT1-related vaccine therapy.
* Patient has a known hypersensitivity to any of the components of the study drug.
* Patient is a staff member of the sponsor or clinical site and is involved in the conduct of the study or the relative of such a staff member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2012-07-31 (Actual); Primary Completion 2017-05-17 (Actual); Study Completion 2017-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vice President Clinical Development and Medical Affairs, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (6):
- United States (6):
  - The University of Arizona Cancer Center - North Campus, Tucson, Arizona
  - UC San Diego Moores Cancer Center, La Jolla, California
  - The University of Chicago Medical Center, Chicago, Illinois
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - The University of Texas, MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- [Derived] Fu S, Piccioni DE, Liu H, Lukas RV, Kesari S, Aregawi D, Hong DS, Yamaguchi K, Whicher K, Zhang Y, Chen YL, Poola N, Eddy J, Blum D. A phase I study of the WT2725 dosing emulsion in patients with advanced malignancies. Sci Rep. 2021 Nov 16;11(1):22355. doi: 10.1038/s41598-021-01707-3. PMID 34785698

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: please note that there were two subjects that never received study drug medication
Groups:
- WT2725 0.3 mg; WT2725 0.9 mg; WT2725 3.0 mg; WT2725 9 mg; WT2725 18 mg; WT2725 27 mg: WT2725; injection WT2725: WT2725 injection Study drug will be administered every 1-4 weeks
Period: Overall Study
Arm/Group | WT2725 0.3 mg | WT2725 0.9 mg | WT2725 3.0 mg | WT2725 9 mg | WT2725 18 mg | WT2725 27 mg
Started | 5 | 5 | 6 | 28 | 9 | 9
Completed | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 5 | 5 | 6 | 28 | 9 | 9
Not completed — Adverse Event | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1 | 13 | 3 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 1 | 3 | 3 | 3
Not completed — progression/treatment failure | 2 | 4 | 3 | 7 | 3 | 5
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0
Not completed — study stopped by sponsor | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | WT2725 0.3 mg | WT2725 0.9 mg | WT2725 3.0 mg | WT2725 9 mg | WT2725 18 mg | WT2725 27 mg | Total
Number analyzed (Participants) | 5 | 5 | 6 | 28 | 9 | 9 | 62
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 3 | 4 | 15 | 7 | 5 | 38
  >=65 years | 1 | 2 | 2 | 13 | 2 | 4 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.4 (8.96) | 62.6 (7.99) | 63.0 (9.25) | 57.5 (15.46) | 51.3 (16.14) | 59.4 (15.83) | 58.0 (14.17)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 6 | 17 | 2 | 1 | 33
  Male | 1 | 2 | 0 | 11 | 7 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 0 | 0 | 4
  Not Hispanic or Latino | 4 | 4 | 5 | 27 | 9 | 8 | 57
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 1 | 1 | 0 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 1 | 0 | 1 | 1 | 0 | 4
  White | 3 | 3 | 5 | 27 | 8 | 7 | 53
  More than one race | 1 | 0 | 0 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 6 | 28 | 9 | 9 | 62
ECOG Performance Status [n(%)] The Eastern Cooperative Oncology Group (ECOG) score [Count of Participants; unit: Participants] — Grade Performance Status 0 Fully active, able to carry on all pre-disease performance without restriction
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, eg, light house work, office work
  2. Ambulatory and capable of all self care but unable to carry out any work activities. Up and about more than 50% of waking hours
  3. Capable of only limited self care, confined to bed or chair more than 50% of waking hours
  4. Completely disabled. Cannot carry on any self care. Totally confined to bed or chair
  5. Dead
  Participants
    0 | 1 | 2 | 6 | 11 | 1 | 3 | 24
    1 | 4 | 3 | 0 | 16 | 8 | 5 | 36
    2 | 0 | 0 | 0 | 1 | 0 | 1 | 2
    3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
    4 | 0 | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Occurrence of Dose-limiting Toxicities and Adverse Events
Description: Evaluation of the safety and tolerability of WT2725 Dosing Emulsion based on the occurrence of DLT and AEs The safety and tolerability of WT2725 Dosing Emulsion will be evaluated based on the occurrence of DLT and AEs, and the findings from clinical laboratory tests, vital signs measurements, body weight measurements, and electrocardiogram (ECG) results. The incidence of DLT will be evaluated during the DLT Evaluation Period, which extends from the day of the first dose to just prior to the fifth dose of study drug (Days 1 to 29). No more than 4 doses of study drug will be administered during the DLT Evaluation Period.
Time Frame: Up to 4 months
Population: Safety Population (defined as all enrolled patients who received at least one dose of study drug.)
Measure: Number; unit: number of occurances
Arm/Group | WT2725 0.3 mg | WT2725 0.9 mg | WT2725 3.0 mg | WT2725 9 mg | WT2725 18 mg | WT2725 27 mg
Number analyzed (Participants) | 5 | 5 | 6 | 28 | 9 | 9
number of occurances | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD) of WT2725 Based on the Evaluation of Dose-limiting Toxicity (DLT)
Time Frame: Day 1 - Day 29
Population: Safety Population (defined as all enrolled patients who received at least one dose of study drug.)
Measure: Number; unit: Dose Limiting Toxicity
Arm/Group | WT2725 0.3 mg | WT2725 0.9 mg | WT2725 3.0 mg | WT2725 9 mg | WT2725 18 mg | WT2725 27 mg
Number analyzed (Participants) | 5 | 5 | 6 | 28 | 9 | 9
Dose Limiting Toxicity | 0 | 0 | 0 | 0 | 0 | 0
Statistical Analysis 1: Comparison: WT2725 0.3 mg vs WT2725 0.9 mg vs WT2725 3.0 mg vs WT2725 9 mg vs WT2725 18 mg vs WT2725 27 mg; The MTD could not be established for this study as no DLTs occurred at doses up to and including 27.0 mg; Test type: Other — None specified; The MTD could not be established for this study as no DLTs occurred at doses up to and including 27.0 mg

3. Secondary Outcome: Antitumor Responses to WT2725 Based on the Immune-related Response Criteria (irRC)
Description: Tumor response, as evaluated according to irRC, was based on total measurable tumor burden in patients with solid tumors (ie, non-AML patients). Tumor assessments will be conducted during screening, and then every 8 weeks after the first dose of study drug. All tumor assessments may be performed within ±7 days of the scheduled assessment. All patients should complete an End of Study visit within 28 days after the last dose of study drug and prior to the start of alternate antineoplastic therapy.
Time Frame: Day 1 - within 28 days after last dose
Population: Efficacy irRC population: including all the patients in the Safety population who are not AML patients and whose lesions are measureable and have at least one posttreatment assessment.
Measure: Number; unit: participants
Arm/Group | WT2725 0.3 mg | WT2725 0.9 mg | WT2725 3.0 mg | WT2725 9 mg | WT2725 18 mg | WT2725 27 mg
Number analyzed (Participants) | 4 | 4 | 6 | 18 | 3 | 5
participants | 0 | 0 | 0 | 2 | 0 | 1

4. Secondary Outcome: Immune Response to WT2725
Description: The modified IWG response criteria were used to assess drug activity in AML patients. Tumor assessments will be conducted during screening, and then every 8 weeks after the first dose of study drug. All tumor assessments may be performed within ±7 days of the scheduled assessment. All patients should complete an End of Study visit within 28 days after the last dose of study drug and prior to the start of alternate antineoplastic therapy.
Time Frame: Day 1 - within 28 days after last dose
Population: Efficacy population for modified IWG response: includes all the AML patients in the Safety population who have >5% marrow blasts or >50 copy/μｇRNA of quantitative RT-PCR for WT1 transcript before the first date/time of study drug and who have at least one posttreatment assessment.
Measure: Number; unit: participants
Arm/Group | WT2725 0.3 mg | WT2725 0.9 mg | WT2725 3.0 mg | WT2725 9 mg | WT2725 18 mg | WT2725 27 mg
Number analyzed (Participants) | 0 | 0 | 0 | 5 | 3 | 1
participants |  |  |  | 3 | 2 | 0

ADVERSE EVENTS:
Time Frame: One month
Description: Serious adverse events (SAEs) will be defined as: • AEs that occurred on or after the first dose of study drug and on or before the 30th day after the last dose of study drug, • AEs with a missing start date and a stop date on or after the first dose of study drug, or • AEs with both a missing start and stop date.
Arm/Group | WT2725 0.3 mg | WT2725 0.9 mg | WT2725 3.0 mg | WT2725 9 mg | WT2725 18 mg | WT2725 27 mg
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/28 | 0/9 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 1/6 | 8/28 | 3/9 | 5/9
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5 | 0/6 | 0/28 | 0/9 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | WT2725 0.3 mg (N=5) | WT2725 0.9 mg (N=5) | WT2725 3.0 mg (N=6) | WT2725 9 mg (N=28) | WT2725 18 mg (N=9) | WT2725 27 mg (N=9)
Bacteraemia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Eye infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Parainfluenzae virus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Viral sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tumor necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Mental Status Changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillar hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash maculopapular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (3):
  • Study Protocol: Final Protocol (2014-12-03): https://cdn.clinicaltrials.gov/large-docs/42/NCT01621542/Prot_000.pdf
  • Study Protocol: Amendment history (2016-08-31): https://cdn.clinicaltrials.gov/large-docs/42/NCT01621542/Prot_001.pdf
  • Statistical Analysis Plan (2017-10-21): https://cdn.clinicaltrials.gov/large-docs/42/NCT01621542/SAP_002.pdf